CLINICAL TRIAL: NCT05133739
Title: A Randomized, Blinded Evaluator, Multicenter, Prospective, Between-subjects Clinical Study to Evaluate Safety and Effectiveness of RHA®4 for the Treatment of Midface Volume Deficiency
Brief Title: RHA®4 for Midface Volume Deficiency
Status: Completed | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-RHA-2004
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Cheek Augmentation; Correction of Age-related Midface Contour Deficiencies
Keywords: Dermal filler; Hyaluronic Acid; Midface; Cannula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded-Live Evaluator
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- RHA®4 (Experimental)
  Interventions: Device: injection of RHA®4 in Midface
- Comparator Device (Active Comparator)
  Interventions: Device: injection of Comparator Product in Midface

INTERVENTIONS:
Device: injection of RHA®4 in Midface — RHA® 4 is a sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer.
  Up to 3.0 mL injected per cheek (subcutaneous and/or supraperiosteal layer). Touch-up treatment provided at 4 weeks (up to 3.0 mL per cheek).
  Arms: RHA®4
Device: injection of Comparator Product in Midface — Comparator product is sterile, biodegradable, colorless gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE.
  Up to 3.0 mL injected per cheek (subcutaneous and/or supraperiosteal layer). Touch-up treatment provided at 4 weeks (up to 3.0 mL per cheek).
  Arms: Comparator Device

SUMMARY:
This is a prospective, randomized, controlled, blinded evaluator, multicenter, between subjects clinical study to identify whether RHA4 is non-inferior to a comparator device for treatment of midface volume deficiency 8 weeks after the last treatment (initial or touch-up).

At Screening, the treating investigator (TI) and the Blinded Live Evaluator (BLE) will evaluate independently the subject's midface using the validated 5-grade Teoxane Midface Volume Deficit Scale (TMVDS) for eligibility of the subject for the study. The BLE will establish a pretreatment score for assessment of effectiveness.

If the assessments of the TI and the BLE are the same or differ exactly by 1 point of the scale, the difference will be considered acceptable. The TI and the BLE need to agree that the subject meets the eligibility criterion (TMVDS grade 2 to 3). If the subject is eligible, the BLE's assessment will be used for the Baseline of the primary endpoint.

Eligible subjects will be enrolled and randomly assigned in a 3:1 ratio at Screening to receive RHA4 or comparator product.

The TI will administer the fillers, and if necessary, subjects will receive a touch-up treatment with the same product that they received on Visit 1, 4 weeks after the initial treatment to optimize the results. If the touch-up treatment is administered, the subject will be asked to come to the site for an additional visit 4 weeks after the touch-up injection.

Subjects will be followed for 52 weeks after their last treatment (initial treatment or touch-up), at which point, they will be offered re-treatment with RHA® 4, regardless of their original treatment, provided that the TI deems the treatment to be appropriate and the subject agrees. Reasons for not administering the re-treatment will be documented.

The subject will then be followed for an additional 12 weeks before exiting the study. If the subject or the TI declines re-treatment, this visit (52 weeks after the last treatment) will be considered the study Exit visit.

For subjects with re-treatment, the Exit visit will be 12 weeks after the re-treatment.

The TI will conduct safety and effectiveness evaluations at each study visit, which will occur: at 4 weeks after the initial and touch-up treatment, 8, 24, and 52 weeks after the last treatment, and after re treatment or until all treatment-related ongoing adverse events (AEs) have resolved or resolved with sequelae as per TI judgment or if follow-up is no longer possible.

A follow-up telephone call for safety will be performed 3 days after each treatment.

Subjects will report their common treatment responses (CTRs) in a subject diary for 30 days after each injection. The diary will also include a list of selected AEs potentially associated with injection of dermal fillers for subjects to report if applicable. All efforts should be made by the TI to schedule the applicable visits to allow completion of the CTR diary.

A BLE will conduct assessments of effectiveness during the study, including assessment of the primary endpoint 8 weeks after the last treatment.

The BLE will be blinded to allocation to groups (RHA4 group or comparator product group).

Furthermore, to ensure that they remain blinded and unbiased when making their assessments throughout the study, the BLE, TI, and subjects will not be allowed to refer to each other's effectiveness assessments. All subjects will be instructed to not discuss their study treatment, AEs, or CTRs with the BLE.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older
* Female subjects of childbearing potential must have a negative UPT and practice a reliable method of contraception throughout the study.
* Seeking treatment of midface volume deficiency (realistic and achievable as per TI opinion)
* Having midface volume loss of grades 2 to 3 on the TMVDS (ranging from 0 = absent to 4 = very severe). The BLE and TI must independently assess and agree that this criterion is met; however, concordance of fullness is not required. If the assessments of the TI and the BLE are the same or differ by exactly 1 point on the scale, this difference is considered acceptable. If the assessments differ by 2 points or more on the scale, the subject will not be eligible.
* Having cheeks of the same TMVDS grade on the left and right side of the face (i.e., approximate bilateral symmetry)
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Sign the IRB-approved ICF, Photographic Release Form and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study- related procedures being performed.

Exclusion Criteria:

* Known hypersensitivity or previous allergic reaction to any component of the study devices.
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
* History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
* History of connective tissue disease.
* Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
* Exposure to any other investigational drug/device within 90 days of entering the study or planning to participate in another investigation during the course of the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- United States, Massachusetts, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RHA®4 | Comparator Device
Started | 152 | 49
ITT Population | 152 | 49
PP Population | 131 | 42
Completed | 126 | 43
Not Completed | 26 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RHA®4 | Comparator Device | Total
Number analyzed (Participants) | 152 | 49 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (9.97) | 55.6 (7.85) | 55.5 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 46 | 180
  Male | 18 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 6 | 24
  White | 130 | 42 | 172
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 152 | 49 | 201
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type as determined by the Treating Investigator on the skin tone scale developed to classify skin coloring and response to ultraviolet (UV) radiation. The scale contains 6 grades:
  I: Pale white skin; Always burns, does not tan. II: Fair skin; Burns easily, tans poorly. III: Darker white skin; Tans after initial burn. IV: Light brown skin; Burns minimally, tans easily. V: Brown skin; Rarely burns, tans darkly easily. VI: Dark brown or black skin; Never burns, always tans darkly.
  Participants
    Type I-III | 107 | 36 | 143
    Type IV-VI | 45 | 13 | 58

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of RHA®4 to the Change From Baseline for Subjects Treated With Comparator Product at 8 Weeks After the Last Treatment as Assessed by the BLE Using the Teoxane Midface Volume Deficit Scale (TMVDS).
Description: A change in the TMVDS ≥1 grade compared to pretreatment will be considered clinically meaningful.
  In order to confirm sensitivity 8 weeks after the last treatment: the proportion of responders with a ≥1-grade point on the TMVDS scale for Comparator product 8 weeks after the last treatment when compared to Baseline must be ≥70%.
  The TMVDS is a validated 5-point scale for assessing midface volume deficit. Possible scores range from 0 (Absent) to 4 (Very Severe).
Time Frame: 8 weeks after the last treatment
Population: Primary endpoint on the PP population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 131 | 42
score on a scale | -1.3 (0.80) | -1.3 (0.65)

2. Secondary Outcome: Change From Baseline in TMVDS Score as Assessed by the BLE at 24 and 52 Weeks After Last Treatment,and Weeks After Re-treatment if Applicable.
Description: A change in the TMVDS ≥1 grade compared to pre-treatment will be considered clinically meaningful.
  The TMVDS is a validated 5-point static scale for assessing midface volume deficit. Possible scores range from 0 (Absent) to 4 (Very Severe).
Time Frame: Week 24, 52 after last treatment, week 12 after re-treatment
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 152 | 49
score on a scale
  Week 24 after last treatment: number analyzed (Participants) | 130 | 44
  Week 24 after last treatment | -1.1 (0.79) | -1.0 (0.76)
  Week 52 after last treatment: number analyzed (Participants) | 128 | 44
  Week 52 after last treatment | -0.9 (0.79) | -0.8 (0.69)
  Re-treatment: 12 weeks post re-treatment: number analyzed (Participants) | 75 | 28
  Re-treatment: 12 weeks post re-treatment | -1.1 (0.91) | -1.2 (0.69)

3. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the BLE.
Description: he Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
Time Frame: Week 8, 24, 52 after last treatment, week 12 after re-treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 152 | 49
Participants
  Week 8 after last treatment: number analyzed (Participants) | 137 | 45
  Week 8 after last treatment | 129 | 44
  Week 24 after last treatment: number analyzed (Participants) | 130 | 44
  Week 24 after last treatment | 111 | 37
  Week 52 after last treatment: number analyzed (Participants) | 128 | 44
  Week 52 after last treatment | 97 | 30
  Re-treatment: 12 weeks post re-treatment: number analyzed (Participants) | 75 | 28
  Re-treatment: 12 weeks post re-treatment | 63 | 26

4. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the "Satisfaction With Cheeks" FACE-Q Scale Questionnaire at Each Visit, at Rest.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 5 questions with a score linked to answers (1 being "Very Dissatisfied" and 4 being "Very Satisfied").
  To calculate the FACE-Q score, outcomes from all 5 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
Time Frame: Change from Baseline at Weeks 8, 24, 52 after last treatment,12 weeks after re-treatment
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 152 | 49
score on a scale
  Week 8 after last treatment: number analyzed (Participants) | 137 | 45
  Week 8 after last treatment | 53.0 (27.15) | 49.5 (27.20)
  Week 24 after last treatment: number analyzed (Participants) | 131 | 44
  Week 24 after last treatment | 48.0 (27.65) | 52.5 (23.48)
  Week 52 after last treatment: number analyzed (Participants) | 128 | 44
  Week 52 after last treatment | 38.6 (28.85) | 38.1 (31.07)
  Re-treatment: 12 weeks post re-treatment: number analyzed (Participants) | 75 | 28
  Re-treatment: 12 weeks post re-treatment | 50.8 (29.97) | 59.3 (21.76)

5. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the "Satisfaction With Cheeks" FACE-Q Scale Questionnaire at Each Visit, When Smiling
Description: as for outcome 4
Time Frame: Change from Baseline at Weeks 8, 24, 52 after last treatment and 12 week after re-treatment.
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 152 | 49
score on a scale
  Week 8 after last treatment: number analyzed (Participants) | 137 | 45
  Week 8 after last treatment | 56.1 (27.67) | 51.3 (29.79)
  Week 24 after last treatment: number analyzed (Participants) | 131 | 44
  Week 24 after last treatment | 49.5 (29.33) | 53.2 (26.68)
  Week 52 after last treatment: number analyzed (Participants) | 128 | 44
  Week 52 after last treatment | 39.6 (29.78) | 41.5 (31.84)
  Re-treatment: 12 weeks post re-treatment: number analyzed (Participants) | 75 | 28
  Re-treatment: 12 weeks post re-treatment | 53.1 (28.43) | 58.2 (21.87)

6. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at Weeks 8, 24, 52 After Last Treatment and 12 Weeks After Re-treatment.
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
Time Frame: Week 8, 24, 52 after last treatment, week 12 after re-treatment
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 | Comparator Device
Number analyzed (Participants) | 152 | 49
Participants
  Week 8 after last treatment: number analyzed (Participants) | 137 | 45
  Week 8 after last treatment | 123 | 43
  Week 24 after last treatment: number analyzed (Participants) | 131 | 44
  Week 24 after last treatment | 119 | 39
  Week 52 after last treatment: number analyzed (Participants) | 128 | 44
  Week 52 after last treatment | 106 | 38
  Re-treatment: 12 weeks post re-treatment: number analyzed (Participants) | 75 | 28
  Re-treatment: 12 weeks post re-treatment | 73 | 28

ADVERSE EVENTS:
Time Frame: 52 to 64 (for patients receiving re-treatment) weeks
Arm/Group | RHA®4 | Comparator Device
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/152 | 3/49
Other Adverse Events (participants affected / at risk) | 36/152 | 8/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA®4 (N=152) | Comparator Device (N=49)
COMPLICATIONS FROM HERNIA REPAIR SURGERY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — not related to study device or study procedure
COVID-19 INFECTION (Infections and infestations) | 1 (1) | 0 (0) — Not related to the study device or study procedure
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) — Not related to the study device or study procedure
P16 POSITIVE OROPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Not related to the study device or study procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHA®4 (N=152) | Comparator Device (N=49)
Injection Site Mass (General disorders) | 17 | 3
Injection Site Induration (General disorders) | 8 | 5
Injection Site Pain (General disorders) | 5 | 1
Injection Site Discoloration (General disorders) | 5 | 0
Headache (Nervous system disorders) | 21 | 5
Covid-19 (Infections and infestations) | 9 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT05133739/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05133739/SAP_001.pdf